CLINICAL TRIAL: NCT02257801
Title: Effects of Lutein on Learning and Memory in Chronically Stressed Subjects and in an Acute Stressful Situation (TSST - Trier Social Stress Test): A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Lutein on Learning and Memory in Chronically Stressed Subjects and in an Acute Stressful Situation (TSST - Trier Social Stress Test): A Randomized, Double-blind, Placebo-controlled Trial)
Acronym: MemLearn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-11-02-LUTE / D1-2011
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Healthy But Chronically Stressed
Keywords: Memory; Cognition; Execute Function; Attention; Mood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nutritional beverage fortified with 6mg lutein/day (Experimental)
  Interventions: Dietary Supplement: Nutritional beverage fortified with 6mg lutein/day
- Nutritional beverage fortified with 12mg lutein/day (Experimental)
  Interventions: Dietary Supplement: Nutritional beverage fortified with 12mg lutein/day
- Nutritional beverage fortified with 0mg lutein/day (Placebo Comparator)
  Interventions: Dietary Supplement: Nutritional beverage fortified with 12mg lutein/day

INTERVENTIONS:
Dietary Supplement: Nutritional beverage fortified with 6mg lutein/day — 2 beverages (each containing 3mg lutein) per day (total of 6mg lutein/day) for a total of 4 months
  Arms: Nutritional beverage fortified with 6mg lutein/day
Dietary Supplement: Nutritional beverage fortified with 12mg lutein/day — 2 beverages (each containing 6mg lutein) per day (total 12mg lutein/day) for a total of 4 months
  Arms: Nutritional beverage fortified with 12mg lutein/day
Dietary Supplement: Nutritional beverage fortified with 12mg lutein/day — 2 beverages (each containing 0mg lutein) per day (total 0mg lutein/day) for a total of 4 months
  Arms: Nutritional beverage fortified with 0mg lutein/day

SUMMARY:
The purpose of this study is to study effects of a four months lutein supplementation (in form of a lutein fortified nutritional beverage) on general learning and memory performance as well as on acute stress-induced changes in learning and memory performance in chronically stressed males and females using 2 different lutein doses in comparison to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 50 - 70 yrs
* Subjects perceiving themselves as chronically stressed and as verified by the TICS questionnaire with scores > 18 and < 48.
* Subject is willing to maintain his or her habitual diet and physical activity patterns throughout the study period
* Subject has a body mass index (BMI) of ≥ 18.50 and ≤ 32.00 kg/m2 at screening.
* Subject is willing to abstain from consuming alcoholic drinks 24 h and from consuming caffeine and caffeine containing products 12 h prior to test days until the end of each visit
* Subject is willing to refrain from heavy physical activity 12 h prior to test days
* Subject finds the taste of the nutritional drink acceptable and is willing to consume 2 drinks per day for the whole study duration
* Subject understands the study procedures and signs the informed consent to participate in the study

Exclusion Criteria:

* Subject has a positive drug screening of amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, opiates, phencyclidine or tricyclic antidepressants at screening or at any of the admission days
* Subject has a positive breath alcohol (as a test for alcohol consumption) or breath carbon monoxide (as test for smoking habits and to exclude smokers) at screening or at any of the admission days
* Subject has any health conditions that would prevent from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the Investigator on the basis of medical history and routine laboratory test results
* Subjects with a history of renal or hepatic disease that is likely to interfere with the metabolism or excretion of the test product
* Subject has donated more than 300 mL of blood during the last three months prior to screening
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mm Hg) at screening
* Subject has a history of psychological illness or condition that interferes with the subject's ability to understand the requirements of the study
* Subject has Diabetes Mellitus
* Subject has a history/ presence of cancer during the last two years (excluding non-melanoma skin cancer)
* Excessive caffeine consumption (>400 mg caffeine/d or ≥4 cups of caffeinated coffee/d), following screening and throughout the study period
* Use of antibiotics or signs of active systemic infections. Treatment visits might be rescheduled
* Subject is on any medication (with the exception of contraception and short-term use of pain treatment e.g. against headache (i.e. 1-2 day use of analgetics such as Paracetamol or ASS) as well as persistent (for at least three months) and well-adjusted medication (e.g. thyroid and blood pressure medication) with no influence on study outcome as judged by the investigator)
* Subject is currently on a regular oral nutrition solution such as Ensure®, Boost® or similar products. Regular is defined as one or more bottles/ cans per day average consumption over the last 10 or more days
* Subjects who are on a significant hypocaloric diet aiming for significant weight loss
* Use of dietary supplements containing any of the following: lutein, ginkgo biloba, St. John's wort, ginseng, gotu kola (Indian pennywort); daily doses of vitamin E (≥30 mg/d) or folic acid (≥400 μg/d); thiamine, riboflavin, and/or pyridoxine (≥2 mg/d); and eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA) or a combination of EPA + DHA (≥500 mg/d) within 2 weeks prior to screening
* Subject is a vegetarian
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 60g (men)/ 40g (women) pure alcohol per day (1.5 l / 1 l beer resp. 0.75 l / 0.5 l wine)
* Subject has a known allergy or sensitivity to the study product or any ingredients of the study product or meals provided, especially against soy and milk protein
* Subject is pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation
* Subject is unable to perform the tests on the CANTAB system during training as being flagged by the software

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visual Memory (Paired Associates Learning (PAL / CANTAB)) | Day 0 (baseline) - day 57
  Visual Memory Task on a computer. Outcome measurements: Change of accuracy (total error adjusted) from baseline measurement to 2 months
Visual Memory (Paired Associates Learning (PAL / CANTAB)) | Day 0 (baseline) - day 113
  Visual Memory Task on a computer. Outcome measurements: Change of accuracy (total error adjusted) from baseline measurement to 4 months
Visual Memory (Verbal Recognition Memory (VRM /CANTAB)) | Day 0 (baseline) - day 57
  Visual Memory Task on a computer. Outcome measurements: Change of accuracy (total number of words correct on immediate recall (the sum of the two free recall trials immediately after each presentation) and delayed recall (the number of correctly recalled words after a delay of approximately 30 min)) from baseline measurement to 2 months
Visual Memory (Verbal Recognition Memory (VRM /CANTAB)) | Day 0 (baseline) - day 113
  Visual Memory Task on a computer. Outcome measurements: Change of accuracy (total number of words correct on immediate recall (the sum of the two free recall trials immediately after each presentation) and delayed recall (the number of correctly recalled words after a delay of approximately 30 min)) from baseline measurement to 4 months
Executive Function (Spatial Working Memory (SWM / CANTAB)) | Day 0 (baseline) - day 57
  Executive Memory Task on a computer. Outcome measurements: Change of accuracy (the total number of between search errors at 4-, 6- and 8-box stages and the strategy score) from baseline measurement to 2 months
Executive Function (Spatial Working Memory (SWM / CANTAB)) | Day 0 (baseline) - day 113
  Executive Memory Task on a computer. Outcome measurements: Change of accuracy (the total number of between search errors at 4-, 6- and 8-box stages and the strategy score) from baseline measurement to 4 months
Executive Function (Spatial Span (SSP / CANTAB)) | Day 0 (baseline) - day 57
  Executive Memory Task on a computer. Outcome measurements: Change of accuracy (Span length forwards) from baseline measurement to 2 months
Executive Function (Spatial Span (SSP / CANTAB)) | Day 0 (baseline) - day 113
  Executive Memory Task on a computer. Outcome measurements: Change of accuracy (Span length forwards) from baseline measurement to 4 months
Attention and Concentration (Reaction Time (RTI / CANTAB)) | Day 0 (baseline) - day 57
  Attention and Concentration Task on a computer. Outcome measurements: Change of reaction time from baseline measurement to 2 months
Attention and Concentration (Reaction Time (RTI / CANTAB)) | Day 0 (baseline) - day 113
  Attention and Concentration Task on a computer. Outcome measurements: Change of reaction time from baseline measurement to 4 months
Attention and Concentration (Rapid Visual Information Processing (RVP / CANTAB)) | Day 0 (baseline) - day 57
  Attention and Concentration Task on a computer. Outcome measurements: Change of target sensitivity and response latency from baseline measurement to 2 months
Attention and Concentration (Rapid Visual Information Processing (RVP / CANTAB)) | Day 0 (baseline) - day 113
  Attention and Concentration Task on a computer. Outcome measurements: Change of target sensitivity and response latency from baseline measurement to 4 months
Verbal Fluency: Regensburg Verbal Fluency Test (RWT) | Day 0 (baseline) - day 57
  Verbal Fluency Task on a computer. Outcome measurements: Change of accuracy (amount of correct answers, breaches of rules, repetitions and total errors) from baseline measurement to 2 months
Verbal Fluency: Regensburg Verbal Fluency Test (RWT) | Day 0 (baseline) - day 113
  Verbal Fluency Task on a computer. Outcome measurements: Change of accuracy (amount of correct answers, breaches of rules, repetitions and total errors) from baseline measurement to 4 months

SECONDARY OUTCOMES:
Visual Memory after TSST (Paired Associates Learning (PAL / CANTAB)) | Day 113
  Visual Memory PAL will be tested before and after an acute social stress test (Trier Social Stress Test (TSST)). Outcome measure: Difference in accuracy (total error adjusted) from before to after TSST.
Visual Memory after TSST (Verbal Recognition Memory (VRM /CANTAB)) | Day 113
  Visual Memory VRM will be tested before and after an acute social stress test (Trier Social Stress Test (TSST)). Outcome measure: Difference in accuracy from before to after TSST.
Executive Function after TSST (Spatial Working Memory (SWM / CANTAB)) | Day 113
  Executive Function SWM will be tested before and after an acute social stress test (Trier Social Stress Test (TSST)). Outcome measure: Difference in accuracy from before to after TSST.
Executive Function after TSST (Spatial Span (SSP / CANTAB)) | Day 113
  Executive Function SSP will be tested before and after an acute social stress test (Trier Social Stress Test (TSST)). Outcome measure: Difference in accuracy from before to after TSST.
Mood (Visual Analog Scale (VAS)) | Day 0 (baseline) to day 57
  Mood will be assessed by VAS. Outcome variables on: alertness, calmness and contentment. Changes of these parameters from baseline day to day 57 and from before to after cognitive test batteries on test days as described above.
Mood (Visual Analog Scale (VAS)) | Day 0 (baseline) to day 113
  Mood will be assessed by VAS. Outcome variables on: alertness, calmness and contentment. Changes of these parameters from baseline day to day 113 and from before to after cognitive test batteries on test days as described above.
Stress (Perceived Stress Scale (PSS)) | Day 0 (baseline) to day 57
  Changes on stress levels will be assessed by PSS. Outcome variables: changes of how unpredictable, uncontrollable, and overloaded subjects perceive their lives.
Stress (Perceived Stress Scale (PSS)) | Day 0 (baseline) to day 113
  Changes on stress levels will be assessed by PSS. Outcome variables: changes of how unpredictable, uncontrollable, and overloaded subjects perceive their lives.
Anxiety (State-Trait-Anxiety Inventory (STAI)) | Day 113
  Changes on personal sensed anxiety levels will be assessed by the STAI questionnaire. Outcome variables: changes of state or trait anxiety scale from before TSST to after the TSST on day 113.
Erythrocyte and serum lutein levels | Day 0 (baseline) to day 113
  Changes in erythrocyte and serum lutein levels will be assessed between baseline and day 113.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Clemens, MD, Principal Investigator — DAaCRO GmbH
Locations (1):
- DAaCRO GmbH, Trier, Trier, Germany